CLINICAL TRIAL: NCT01229358
Title: Prospective, Randomized Clinical Trial of a Silver Eluting Dressing System for Prevention of Lower Extremity Revascularization Wound Complications
Brief Title: Clinical Trial of a Silver Eluting Dressing System
Acronym: SILVER
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other); Michael E. DeBakey VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, C. Keith Ozaki, M.D., F.A.C.S., Associate Professor, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2010-P-001149/1
Record Dates: First submitted 2010-10-26; First posted 2010-10-27 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 2016-01

CONDITIONS: Vascular Disease; Surgery
Keywords: vascular surgery; wound infection; wound complication
MeSH Terms: conditions — Vascular Diseases; Wound Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Silver Eluting Dressing (Experimental): Acticoat Absorbant™ applied as post-operative dressing
  Interventions: Other: Surgical dressing
- Standard Guaze (Active Comparator): Standard dry gauze applied as post-operative dressing
  Interventions: Other: Surgical dressing

INTERVENTIONS:
Other: Surgical dressing — Acticoat Absorbant™ vs standard dry gauze as the immediate post operative dressing
  Other Names: Acticoat Absorbant™, Silver dressing

SUMMARY:
This prospective, multi-institutional randomized clinical trial of a silver ion eluting dressing material compared to standard dry gauze for closed skin incisions after open surgical revascularizations for peripheral vascular occlusive disease. Based on the ability of the silver to lower the bacterial contamination of these vulnerable surgical skin incisions, the investigators hypothesize that immediate application of Acticoat Absorbent® as a post-operative dressing will reduce closed incisional wound complications in patients undergoing lower extremity revascularizations involving infrainguinal skin incisions compared to standard non-silver eluting dressing material.

DETAILED DESCRIPTION:
Rationale:

One of the most common post-operative complications of surgical procedures remains surgical site infection, which causes significant morbidity and healthcare costs (estimated at $1.5 billion per year) among hospitalized patients. Surgical wounds for lower extremity revascularization are particularly prone to infection and dehiscence, with rates in some series as high as 44%(Kent, Bartek et al. 1996). Currently, the Guideline for Prevention of Surgical Site Infection recommends the use of sterile dressing to protect closed incisions for 24 to 48 hour postoperatively. However, no evidence-based recommendations are made with regards to dressing types for use in post-operative incision care.

A plethora of wound dressings are available in the market, with silver-based dressing among these recent innovations. Topical silver treatment is an effective bactericidal agent that does not induce bacterial resistance when used in therapeutic levels. Acticoat Absorbent®(Smith and Nephew, Inc.), an antimicrobial barrier dressing is coated with nanocrystalline silver that delivers a controlled, sustained (up to three days) dose of silver ions. Additionally, this dressing absorbs moisture (minimizing wound maceration), and is safe and effective against a broad range of microorganisms. Acticoat Absorbent® (Acticoat) is indicated for surgical wounds, chronic wounds, and burn wounds; however, data are lacking regarding in its potential role in postoperative surgical incision wound infection prophylaxis.

The Principal Investigator recently completed a non-concurrent, single-institution study of patients who received conventional non-silver containing dressing with Acticoat as post-operative dressing following defined lower extremity revascularizations(Childress, Berceli et al. 2007). The study population comprised 216 patients who underwent 248 cases that met inclusion criteria. Both groups were similar with regards to age at the time of first procedure, gender, race, diabetes, hypertension, current smoking, and renal insufficiency (creatinine >1.5 mg/L). Furthermore, both groups had tissue loss as the most common indication for the lower extremity revascularization procedure, with 47% (55/118) for the control group and 38% (49/130) for the treatment group. Moreover, autogenous vein bypass graft was the most common procedure performed for the control (65/118, 55% of procedures) and treatment (54/130, 42% of procedures) groups.

The surgeons and other providers found the dressing regimen easy to apply and care for post-operatively. Revascularization pulses could be palpated through the dressing, and the low profile permitted identification of post-operative soft tissue changes such as hematomas. Compressive ace bandages could be applied without disturbing the original dressing.

Regarding the primary findings, no substantial dressing material specific complications were noted, including no apparent allergic reactions. The wound complication rate for the control group was 14% (17/118), and for the treatment group was 5% (7/130). Over the intervention phase, the wound overall complication rate fell by 64% (c2 = 5.76, df = 1, p = 0.016).

These findings provide clinical evidence that an Acticoat based dressing system offers a potentially efficacious, cost-effective adjunct to reduce surgical site infections for lower extremity revascularization. Based on this data, we believe that further investigation via multi-center randomized clinical trial is warranted. Thus for the current proposal we hypothesize that immediate application of Acticoat Absorbent® as a post-operative dressing would reduce closed incisional wound complications in patients undergoing lower extremity revascularizations involving infrainguinal skin incisions will result in a clinically significant reduction in wound complication rates compared to standard non-silver eluting dressing material.

Procedure:

* Patient randomized in OR after wound closure completed
* Wound closure technique at the discretion of the surgeon (Dermabond is a dressing and can not be utilized)
* Final OR dressing is test (silver vs standard) dressing, secured per surgeon preference
* Original OR dressing stays in place until gross soiling impairs standard wound hygiene, clinical need to remove, or POD#3, whichever comes first
* Subsequent dressings, wound care at the discretion of providers
* Visual wound checks at least at 2 and 4 weeks (+/- 5 days)

Clinical, economic, patient quality of life, and resource utilization data is then collected at standard clinical encounters

Primary Endpoint: Any wound complication within 30 days

Power and Sample Size Calculations:

* Current endpoint rate at least 25%(Kent, Bartek et al. 1996; Nguyen, Brahmanandam et al. 2007)
* Anticipate 10% absolute (40% relative) wound complication rate reduction(Childress, Berceli et al. 2007)
* Power 0.8
* alpha 0.05
* control event rate of 0.25
* treatment event rate of 0.15
* 1:1 randomization
* -->total study sample size 250 per group (500 total).

ELIGIBILITY:
Inclusion Criteria:

* Adult patient capable of informed consent who completes consent process
* Undergoing open (an incision below inguinal ligament) surgical procedure for peripheral arterial vascular disease in which it is anticipated that the incisions will be closed. Open cases combined with endovascular approaches acceptable.

Exclusion Criteria:

* Age less than 18
* Known allergy to silver or alginate
* Participation in another interventional clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2010-10; Primary Completion 2013-09 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Wound complication | Within 30 days of index procedure
  * No Wound Complication
  * Superficial Incisional SSI: Infection that occurs within 30 days after the operation and infection involves only skin/ SQ tissue of the incision
  * Deep Incisional SSI: Infection that occurs within 30 days after operation and infection appears to be related to the operation and infection involved deep tissues (fascial/muscle layers) of the incision
  * Other (seroma, lymphocele, hematoma, etc)

CONTACTS AND LOCATIONS:
Overall Officials: C Keith Ozaki, MD, Principal Investigator — Brigham and Women's Hospital
Locations (3):
- United States (3):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Michael Debakey Veterans Affairs Medical Center, Houston, Texas

REFERENCES:
- [Background] Childress BB, Berceli SA, Nelson PR, Lee WA, Ozaki CK. Impact of an absorbent silver-eluting dressing system on lower extremity revascularization wound complications. Ann Vasc Surg. 2007 Sep;21(5):598-602. doi: 10.1016/j.avsg.2007.03.024. Epub 2007 May 23. PMID 17521872
- [Background] Nguyen LL, Brahmanandam S, Bandyk DF, Belkin M, Clowes AW, Moneta GL, Conte MS. Female gender and oral anticoagulants are associated with wound complications in lower extremity vein bypass: an analysis of 1404 operations for critical limb ischemia. J Vasc Surg. 2007 Dec;46(6):1191-1197. doi: 10.1016/j.jvs.2007.07.053. PMID 18154995
- [Background] Khuri SF, Daley J, Henderson W, Hur K, Demakis J, Aust JB, Chong V, Fabri PJ, Gibbs JO, Grover F, Hammermeister K, Irvin G 3rd, McDonald G, Passaro E Jr, Phillips L, Scamman F, Spencer J, Stremple JF. The Department of Veterans Affairs' NSQIP: the first national, validated, outcome-based, risk-adjusted, and peer-controlled program for the measurement and enhancement of the quality of surgical care. National VA Surgical Quality Improvement Program. Ann Surg. 1998 Oct;228(4):491-507. doi: 10.1097/00000658-199810000-00006. PMID 9790339
- [Background] Kent KC, Bartek S, Kuntz KM, Anninos E, Skillman JJ. Prospective study of wound complications in continuous infrainguinal incisions after lower limb arterial reconstruction: incidence, risk factors, and cost. Surgery. 1996 Apr;119(4):378-83. doi: 10.1016/s0039-6060(96)80135-8. PMID 8644000
- [Derived] Correia RM, Nakano LC, Vasconcelos V, Cristino MA, Flumignan RL. Prevention of infection in peripheral arterial reconstruction of the lower limb. Cochrane Database Syst Rev. 2025 Oct 29;10(10):CD015022. doi: 10.1002/14651858.CD015022.pub2. PMID 41159585
- [Derived] Ozaki CK, Hamdan AD, Barshes NR, Wyers M, Hevelone ND, Belkin M, Nguyen LL. Prospective, randomized, multi-institutional clinical trial of a silver alginate dressing to reduce lower extremity vascular surgery wound complications. J Vasc Surg. 2015 Feb;61(2):419-427.e1. doi: 10.1016/j.jvs.2014.07.034. Epub 2014 Aug 28. PMID 25175629